CLINICAL TRIAL: NCT01688648
Title: The Comparison of Antiarrhythmic and Myocardial Protective Effect Between Lidocaine, Dexmedetomidine, and Their Combined Infusion in Subjects Undergoing Coronary Artery Bypass Graft
Brief Title: Comparison Between Lidocaine, Dexmedetomidine, and Their Combined Infusion in Subjects Undergoing Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Sung Cho, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2012-07-098-001
Record Dates: First submitted 2012-09-10; First posted 2012-09-20 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Unstable Angina; Coronary Artery Bypass Graft; Dexmedetomidine; Lidocaine; Myocardial Injury; Arrhythmia; Blood Electrolyte Balance
Keywords: Coronary artery bypass graft; dexmedetomidine; lidocaine; myocardial injury; arrhythmia; blood electrolyte balance
MeSH Terms: conditions — Angina, Unstable; Arrhythmias, Cardiac | interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lidocaine group (Experimental): a bolus dose of lidocaine 1.5 mg/kg after anesthetic induction with following lidocaine infusion with 2 mg/kg/hr during the surgery and same dose during postoperative 24 hour in ICU.
  Interventions: Drug: Lidocaine infusion
- Dexmedetomidine group (Experimental): Dexmedetomidine infusion during anesthetic induction with 0.2 mcg/kg/hr followed by 0.3 ~ 0.7 mcg/kg/hr during the surgery
  Interventions: Drug: Dexmedetomidine infusion
- Combined infusion group (Experimental): Combined lidocaine and dexmedetomidine infusion with the dose specified in single infusion group
  Interventions: Drug: Lidocaine infusion; Drug: Dexmedetomidine infusion
- Control group (No Intervention): The group without infusion of lidocaine or dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine infusion — a bolus dose of Lidocaine 1.5 mg/kg after anesthetic induction with following infusion with 2 mg/kg/hr during the surgery and same dose during postoperative 24 hour in ICU.
  Other Names: 2% lidocaine hydrochloride
  Arms: Combined infusion group; Lidocaine group
Drug: Dexmedetomidine infusion — Dexmedetomidine infusion during anesthetic induction with 0.2 mcg/kg/hr followed by 0.3 ~ 0.7 mcg/kg/hr during the surgery
  Other Names: Precedex injection; Dexmedetomidine hydrochloride 118 mcg/ml
  Arms: Combined infusion group; Dexmedetomidine group

SUMMARY:
The aim of the present study is to compare the antiarrhythmic and myocardial protective effect between lidocaine, dexmedetomidine, and their combined infusion in subjects undergoing coronary artery bypass graft.

DETAILED DESCRIPTION:
Lidocaine has been reported to have an antiarrhythmic and myocardial protective effect. A previous study has reported that low-dose lidocaine infusion can decrease the incidence of ventricular fibrillation and tachycardia during the first 24 hours after coronary artery bypass graft (CABG). A recent study also reported that the lidocaine infusion during CABG could decrease the myocardial injury by measuring the CK-MB and Troponin-I blood level.

Dexmedetomidine is an alpha-2 agonist and reduces the sympathetic tone and neuroendocrine stress response. Dexmedetomidine was reported to have a cardioprotective effect by a previous animal study. However, there was no clinical study evaluating the cardioprotective effect of dexmedetomidine.

Therefore, we are trying to evaluate and compare the antiarrhythmic and myocardial protective effect between lidocaine, dexmedetomidine, and their combined infusion in subjects undergoing coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing off-pump coronary artery bypass graft during the study period in Samsung Medical Center

Exclusion Criteria:

* Any patients with plasma aldosterone, or glucocorticoid disorder including primary hyperaldosteronism, renovascular hypertension, rennin-secreting tumor, salt-wasting renal disease, Cushing syndrome
* Patients with recent exogenous steroid administration or previous diuretics therapy
* Patients with recent myocardial infarction
* Those undergoing unplanned cardiopulmonary bypass during the surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Myocardial injury marker | postoperative ICU day 1
  Myocardial injury marker - CK-MB, and Troponin(i) blood level
Myocardial injury marker | postoperative ICU day 2
  Myocardial injury marker - CK-MB, and Troponin(i) blood level
Myocardial injury marker | postoperative ICU day 3
  Myocardial injury marker - CK-MB, and Troponin(i) blood level

SECONDARY OUTCOMES:
The blood sodium, potassium, calcium level | 1 day before surgery day, at the start of anesthetic induction, 2 hour, 4 hour after anesthetic induction, postoperative ICU day 1, 2, 3
  The blood sodium, potassium, calcium level
The incidence of arrhythmia during and after the surgery | 1 day before surgery day, at the start of anesthetic induction, 2 hour, 4 hour after anesthetic induction, postoperative ICU day 1, 2, 3
  The incidence of arrhythmia during and after the surgery:
  Ventricular premature beat,Atrial premature complex, Bigeminy, Trigeminy, Atrial fibrillation, Ventricular tachycardia, Ventricular fibrillation, Atrio-Ventricular block, PSVT, Junctional rhythm, External pacing
Postoperative ICU stay, Hospital stay, Extubation time | 1 day after hospital discharge
  Postoperative ICU stay, Hospital stay
Inotropics use during and after the surgery | 1 day before surgery day, at the start of anesthetic induction, 2 hour, 4 hour after anesthetic induction, , postoperative ICU day 1, 2, 3
  Inotropics and other drug use during and after the surgery: Dopamine, NTG, dobutamine, milrinone, epinephrine, norepinephrine, amiodarone, diltiazem, remifentanil, esmolol, labetalol, nicardipine, Lasix, phenylephrine, lidocaine, sufentanil
The incidence of hypokalemia | 1 day before surgery day, at the start of anesthetic induction, 2 hour, 4 hour after anesthetic induction, , postoperative ICU day 1, 2, 3
  The incidence of hypokalemia

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea